CLINICAL TRIAL: NCT06757205
Title: Analysis of the Personality Characteristics and Lifestyle of Young People Who Access Psychiatric Outpatient Clinics: a Qualitative Study
Brief Title: Analysis of the Personality Characteristics and Lifestyle of Young People Who Access Psychiatric Outpatient Clinics
Acronym: APGP
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7088
Record Dates: First submitted 2024-12-23; First posted 2025-01-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-12

CONDITIONS: Personality; Life Style

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Using a structured questionnaire to collect quantitative and qualitative data on adolescents' experiences and perceptions. The Italian version of the Mentalization Questionnaire (MZQ) was develop — Using a structured questionnaire to collect quantitative and qualitative data on adolescents' experiences and perceptions.
  * The Italian version of the Mentalization Questionnaire (MZQ) was developed as a self-rated instrument to assess mentalization. It consists of 15 items with responses ranging from 1 = 'no agreement at all' to 5 = 'total agreement' on a 5-point Likert scale. Calculated sum scores for the total scale range from 15 to 75 with higher scores indicating lower mentalization capacities.
  * The Toronto Alexithymia Scale (TAS) is a measure of deficiency in understanding, processing, or describing emotions (alexithymia). It has twenty statements rated on a five-point Likert scale. The total score ranges from 40 to 200 and the higher score indicates a greater level of alexithymia.

SUMMARY:
Considering the growing importance of services psychiatric and psychological for adolescence and adulthood incidence of discomfort expressed in this age group, comes assessed the need to provide adequate and targeted services.

Reasons:

The study aims to evaluate the characteristics and trends of adolescents who access the service, in order to frame the type of discomfort expressed and the expectations with respect to access to the service and the resource base on which it can the therapeutic intervention must be thought out and organised. Furthermore, the study aims to identify the factors that influence the request for help and evaluate the quality of the assistance received, with the aim of improving it effectiveness.

ELIGIBILITY:
Inclusion criteria:

- Participants will be selected based on their age between 13 and 21, their availability to sign the informed consent.

Exclusion criteria:

* Patients who do not give their consent are excluded from the study.
* Patients who do not speak fluent Italian or those who due to cognitive and/or thinking characteristics would not be able to understand or complete the questionnaire are also excluded.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study involves the enrollment of 115 adolescents aged between 13-21 years treated at the psychiatric clinic.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Analyze the characteristics of adolescents who access the clinic, both with respect to the discomfort presented and the resources available to them | one year
  Data analysis through qualitative methods to identify recurring trends and patterns.

SECONDARY OUTCOMES:
Relate these characteristics to the ways of relating within the family, through meetings that also involve their parents | one year
  Administration of psychometric scales:
  * The Italian version of the Mentalization Questionnaire (MZQ) was developed as a self-rated instrument to assess mentalization. It consists of 15 items with responses ranging from 1 = 'no agreement at all' to 5 = 'total agreement' on a 5-point Likert scale. Calculated sum scores for the total scale range from 15 to 75 with higher scores indicating lower mentalization capacities.
  * The Toronto Alexithymia Scale (TAS) is a measure of deficiency in understanding, processing, or describing emotions (alexithymia). It has twenty statements rated on a five-point Likert scale. The total score ranges from 40 to 200 and the higher score indicates a greater level of alexithymia.

OTHER OUTCOMES:
Collect useful information to improve the effectiveness and variety of therapeutic paths to be offered to adolescents who consult the clinic and their parents. | one year
  Administration of psychometric scales:
  * The Italian version of the Mentalization Questionnaire (MZQ) was developed as a self-rated instrument to assess mentalization. It consists of 15 items with responses ranging from 1 = 'no agreement at all' to 5 = 'total agreement' on a 5-point Likert scale. Calculated sum scores for the total scale range from 15 to 75 with higher scores indicating lower mentalization capacities.
  * The Toronto Alexithymia Scale (TAS) is a measure of deficiency in understanding, processing, or describing emotions (alexithymia). It has twenty statements rated on a five-point Likert scale. The total score ranges from 40 to 200 and the higher score indicates a greater level of alexithymia.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Mazza, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome, ROMA, Italy

IPD SHARING:
Plan to Share IPD: No